CLINICAL TRIAL: NCT04871620
Title: Reliability of a New Pulse Contour Technique for Diagnosing an Increase in Stroke Volume During a Fluid Challenge for Hemodynamic Optimization in Patients Scheduled for High-risk Abdominal Surgery: Comparison With Transthoracic Echocardiography: COMPARE Study
Acronym: COMPARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/PC-01
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Surgery; Cardiac Output, Low
Keywords: High risk abdominal surgery; hemodynamic optimization; stroke volume; pulse contour
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodynamic optimization: Patients scheduled for intermediate and high-risk abdominal surgery were eligible to participate
  Interventions: Diagnostic Test: >15% SV increase during fluid challenge

INTERVENTIONS:
Diagnostic Test: >15% SV increase during fluid challenge — The stroke volume will be measured before and after 15 minutes fluid challenge with crystalloids

SUMMARY:
The present study aims at assessing the ability of a new pulse contour device for diagnosing a >15% stroke volume (SV) increase during patient hemodynamic optimization by fluid challenge in high risk abdominal surgery.

DETAILED DESCRIPTION:
In European countries, day-7 mortality rate could reach 1-5. %. Emergency conditions, American Society Assessment (ASA) and major surgery were associated with a higher risk of immediate mortality. Moreover, hemodynamic instability is well known to lead to postoperative complications and a higher risk of mortality.

Since, nearly 30 years, optimization of hemodynamic conditions, especially via an optimization of the fluid administration has been shown to improve immediate and long-term patient outcome. This strategy is currently widely accepted and recommended in medium and high-risk surgery. Therefore, optimizing cardiac output and one of its surrogate is proposed over intraoperative surgery. For assessing the cardiac output or the indexed stroke volume, esophageal Doppler and pulse contour technique have been proposed and have shown that they could improve patient outcome.

However, the reliability of esophageal Doppler, pulse contour and non-invasive techniques assessing cardiac output and its ability to detect a change in the initial value of CO have been challenged. Initially, the reliability of a technique for measuring CO has been described by using a correlation coefficient and by building Bland & Altman diagram. However, searching a correlation between two different techniques measuring the same parameter will lead to a correlation. In the same, Bland & Altman technique shows the mean difference between measurements of the same parameters; However, demonstrating a good reliability should be shown by a narrow limit of agreement with no definition of the narrowness. Indeed, a value of cardiac index (CI) = 3 l/min/m2 with a mean difference of 0 +/- 1.1 /min/m2 by Bland & Altman technique mean that the CI value could be within 1 and 5 l/min/m2 that could lead to different treatment such as fluid challenge, vasopressor or inotrope infusion.

An interesting method for comparing two techniques measuring the same parameter could be to challenge one technique versus the other one in decision-making. Applying this method to techniques measuring CO, we could search for the interest of a new technique for diagnosing an increase in CO after a fluid challenge for optimizing cardiac preload and hemodynamic status. Esophageal Doppler is classically recommended for optimizing hemodynamic patient in high-risk surgery.

A new device using pulse contour technology has been available since a few years. Therefore, the present study aims at assessing the ability of this device for diagnosing an increase in CO > 15% during patient hemodynamic optimization by fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ASA status 1-3 who were orally informed and did refuse to participate.
* Patient in whom general anesthesia with tracheal intubation were planned.
* Patient in whom an arterial catheter and a monitoring of cardiac output by esophageal Doppler were indicated for hemodynamic optimization
* Patient with cardiac sinusal mode

Exclusion Criteria:

* Patient < 18-year-old
* Cardiac arrythmia
* Patient with anomaly in oro-pharyngo-esophageal tractus
* Patients with hemostasis anomaly (PT < 30%, platelets < 50 000 elements/mm3)
* Patient in whom the cardiac output monitoring or measurement was not possible by Esophageal Doppler or echography
* Patients in whom cardiac arrythmia occurred during the procedure of hemodynamic optimization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for intermediate and high-risk abdominal surgery were eligible to participate
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Ability of pulse contour for diagnosing a >15% increase in stroke volume | 15 minutes
  Ability of pulse contour for diagnosing a >15% increase in stroke volume

SECONDARY OUTCOMES:
Comparison with the ability of other techniques | 15 minutes
  Comparison with the ability of other techniques (Esophagial Doppler, other pulse contour techniques for diagnosing a >15% SV increase)
Ability for predicting a >15% SV increase | 15 minutes
  Ability of Esophagial Doppler and Pulse contour techniques for predicting a >15% SV increase after rapid infusion of 100ml cristalloid over one minute (mini-fluid challenge)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No